CLINICAL TRIAL: NCT00580983
Title: Optimized Intensity Modulated Irradiation for Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2-21; HUM 43020 Legacy 2002-513 (Other: University of Michigan IRBMED)
Record Dates: First submitted 2007-12-25; First posted 2007-12-27 (Estimated); Results first posted 2014-11-14 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-07

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Paclitaxel; Carboplatin; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemo-IMRT (Experimental): Chemotherapy:
  Chemotherapy will consist of Paclitaxel 30mg/m² IV over 1 hour, followed by Carboplatin (AUC 1) IV over 30 minutes, or Carboplatin 100mg/m² per IV over 30 minutes or Cisplatin 100mg/m² per IV over 1 hour, or Cisplatin (80mg/m²) or Carboplatin (AUC 5) IV on day 1 and 5-Fluorouracil (1000mg/m²) as a 24-hour continuous infusion, daily x 4 days.
  Intensity-modulated Radiation Therapy (IMRT):
  Primary RT: 70 Gy to gross disease and 56-63 Gy to subclinical disease in 35 fractions.
  Post-operative RT: 64 Gy to high-risk targets (postoperative tumor bed, first-echelon nodes) and 57.6 Gy to low-risk targets, in 32 fractions.
  Interventions: Radiation: IMRT; Drug: Paclitaxel; Drug: Carboplatin; Drug: Cisplatin; Drug: 5-Fluorouracil

INTERVENTIONS:
Radiation: IMRT
Drug: Paclitaxel
Drug: Carboplatin
Drug: Cisplatin
Drug: 5-Fluorouracil

SUMMARY:
The purpose of this study is to test whether the use of advanced radiation therapy delivery techniques can spare a patient's normal tissue, including salivary glands, from radiation. This study is being done to try to reduce radiation side effects, especially mouth dryness, which happens with standard radiation methods. In order to reduce these side effects, other normal tissues may receive a different radiation dose (sometimes more) than what would have been received using standard radiation therapy. A secondary goal of this study is to determine if the type of tumor a patient has can be controlled at least as well (or better) using this advanced radiation therapy delivery technique as it would be if the patient was treated with standard radiation therapy.

DETAILED DESCRIPTION:
Studies show that a dose response relationship in the salivary glands exists and that it may be possible to improve significantly post-radiation xerostomia and quality of life if radiation techniques can be devised that would spare the salivary glands while adequately treating the targets. A new treatment modality (computer-optimized IMRT) facilitates increased sparing of noninvolved tissue, specifically the sparing of both parotid glands, and more conformal high-dose delivery to the bilateral neck targets in patients with head and neck cancer. This study will evaluate the benefits regarding xerostomia-specific and general QOL in patients receiving head and neck RT using this modality. Assessment of swallowing dysfunction and aspiration will be made using videofluoroscopy. In addition, this study will evaluate the pattern of local/regional tumor recurrence, to assess whether sparing both parotid glands may cause tumor recurrence in spared neck areas.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have histologically confirmed invasive cancer of the head and neck.
* Irradiation to both neck sides is required.
* Standard radiation techniques would irradiate most of both parotid glands to a high dose (>50 Gy). Patients with oropharyngeal, oral, nasopharyngeal, hypopharyngeal and advanced laryngeal cancer are expected to fulfill this requirement.
* Patients with resectable disease that is either measurable, evaluable or non-measurable disease (post-operative) will be eligible.
* Karnofsky performance status >60
* Patients receiving or not receiving chemotherapy are eligible.
* All patients must sign an informed consent.
* Pre-treatment laboratory criteria:

  * WBC (White Blood Cell) > 3500/ul, granulocyte > 1500/ul.
  * Platelet count > 100,000/ul.
  * Creatinine clearance > 60 cc/min. to receive cisplatin; creatinine clearance 30-59 cc/min to receive carboplatin.
  * Bilirubin < 1.5 mg% with no evidence of obstructive liver disease.
  * AST (Aspartate Aminotransferase) and ALT (Alanine Aminotransferase) equal to or less than 2.5 x upper limit of normal.

Exclusion Criteria:

* Patients who received past irradiation to the head and neck are not eligible.
* Prior head and neck malignancy or history of other prior non-head and neck malignancy within the past 3 years.
* Prior head and neck radiation or prior chemotherapy.
* Documented evidence of distant metastases.
* Active infection.
* Pregnancy or lactation; patients must use effective contraception during the course of the clinical trial.
* Any medical or psychiatric illness which in the opinion of the principal investigator would compromise the patients ability to tolerate this treatment.
* Patients residing in prison.
* Age < 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2003-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Avraham Eisbruch, M.D., Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 90 participants were enrolled however only 80 started treatment. Only 73 participants completed treatment. 7 did not complete the 12 month post radiation therapy (RT)swallowing studies.
Period: Overall Study
Arm/Group | Chemo-IMRT
Started | 80
Completed | 73
Not Completed | 7
Not completed — Did not complete 12 mon post RT studies | 7

BASELINE CHARACTERISTICS:
Population: 90 patients were enrolled. Only 80 patients were treated and 7 patients did not complete the 12 month post-Radiation Therapy (RT) swallowing studies. Therefore only 73 participants were included in the baseline analysis.
Arm/Group | Chemo-IMRT
Number analyzed (Participants) | 73
Age, Continuous [Median (Full Range); unit: years] | 55 [50 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 65
Tumor Location [Number; unit: participants]
  Tonsil | 35
  Base of Tongue | 38
Gross Tumor Volume [Median (Full Range); unit: mL] | 110 [19 to 378]
T Stage [Number; unit: participants] — The TNM (Classification of Malignant Tumours) staging system is a standard system used to describe and summarize how far a patient's cancer has spread. The T indicates the size of the primary tumor. The numbers 0 through 4 indicate increasing severity.
  participants
    Stage 1 | 9
    Stage 2 | 29
    Stage 3 | 17
    Stage 4 | 18
N Stage [Number; unit: participants] — The TNM staging system is a standard system used to describe and summarize how far a patient's cancer has spread. The T describes the extent of spread to nearby lymph nodes. The numbers 0 through 4 indicate increasing severity.
  participants
    Stage 0 | 6
    Stage 1 | 6
    Stage 2 | 55
    Stage 3 | 6
AJCC Stage [Number; unit: participants] — The AJCC staging system is a classification system developed by the American Joint Committee on Cancer (AJCC) for describing the extent of disease progression in cancer patients.
  The TNM (Tumor, Lymph Node, Metastasis) classifications for cancers of the head and neck vary with location. Once the T, N, and M are determined, they are combined, and an overall stage of 0, I, II, III, IV is assigned.
  participants
    Stage III | 9
    Stage IVA | 58
    Stage IVB | 6
Smoking Status [Number; unit: participants]
  Never Smoked | 26
  Previous Smoker | 31
  Current Smoker | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Grade 0-1 Observer-rated Dysphagia
Description: To objectively assess dysphagia and aspiration in patients receiving dysphagia/aspiration-sparing IMRT concurrent with chemotherapy, the percentage of participants with observer-rated dysphagia was calculated.
Time Frame: 12 months
Population: 90 patients were enrolled. Only 80 patients were treated and 7 patients did not complete the 12 month post-Radiation Therapy (RT) swallowing studies. Therefore only 73 patients were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Chemo-IMRT
Number analyzed (Participants) | 73
percentage of participants | 94

2. Secondary Outcome: The Mean Esophageal Radiotherapy Dose in Patients With Strictures and Without Strictures
Description: To assess the relationships between the mean radiotherapy dose delivered and objectively measured dysphagia.
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: Gray (Gy)
Arm/Group | Chemo-IMRT
Number analyzed (Participants) | 73
Gray (Gy)
  Patients with Strictures (N=5) | 48 (17)
  Patients without strictures (N=68) | 27 (12)

ADVERSE EVENTS:
Description: 90 patients were enrolled. Only 80 patients were treated and 7 patients did not complete the 12 month post-Radiation Therapy (RT) swallowing studies. Therefore only 73 patients were included in the adverse events analysis.
Arm/Group | Chemo-IMRT
Serious Adverse Events (participants affected / at risk) | 26/73
Other Adverse Events (participants affected / at risk) | 0/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemo-IMRT (N=73)
Anxiety (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Dobhoff Tube Complication (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 3
Esophageal Stricture (Gastrointestinal disorders) | 1
Fever (General disorders) | 2
Headache (Nervous system disorders) | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hyperlipedemia (Investigations) | 1
Hypertension (Cardiac disorders) | 1
Increased Mucous Secretions (General disorders) | 1
Induration of Skin (Skin and subcutaneous tissue disorders) | 1
Mental Status Change (Psychiatric disorders) | 3
Mucositis (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 7
Neck Pain (General disorders) | 2
Neck Swelling (General disorders) | 1
Odynophagia (Gastrointestinal disorders) | 1
PEG Tube Complications (Surgical and medical procedures) | 1
Pharyngeal Stenosis (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 7
Poor Oral Intake (Metabolism and nutrition disorders) | 1
Skin Redness (Skin and subcutaneous tissue disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Syncope (Nervous system disorders) | 1
Thrush (Gastrointestinal disorders) | 2
Ulceration of the Mucous Membrane (Gastrointestinal disorders) | 1
Urinary Tract Infection (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Weight Loss (General disorders) | 1

LIMITATIONS AND CAVEATS:
No modeling of observer-rated posttherapy dysphagia was performed because of the small number (four) of patients with greater than, or equal to, Grade 2 after 6 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes